CLINICAL TRIAL: NCT00084370
Title: Molecular Alterations in Human Ovarian Epithelium Induced by Chemopreventive Agents in Patients at Elevated Inherited Risk of Ovarian Cancer: A Controlled Pilot Study in Ovarian Cancer Chemoprevention
Brief Title: Celecoxib in Preventing Cancer in Patients at High Risk for Ovarian Epithelial Cancer Who Are Undergoing Prophylactic Oophorectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Partridge, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000352114; UAB-0134
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Ovarian Cancer
Keywords: ovarian epithelial cancer; BRCA1 mutation carrier; BRCA2 mutation carrier
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Celecoxib; Ovariectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Group I: Patients receive oral celecoxib twice daily for 3 months and then undergo prophylactic oophorectomy.
  Interventions: Drug: celecoxib; Procedure: oophorectomy
- Group II (Experimental): Group II: Patients undergo immediate prophylactic oophorectomy.
  Interventions: Procedure: oophorectomy

INTERVENTIONS:
Drug: celecoxib — Patients receive ora celecoxib twice daily for 3 months prior to prophylactic oophorectomy.
  Arms: Group 1
Procedure: oophorectomy

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of celecoxib before prophylactic oophorectomy may be an effective way to prevent the development of ovarian epithelial cancer.

PURPOSE: A controlled pilot trial to study the effectiveness of celecoxib in preventing cancer in patients at high-risk for ovarian epithelial cancer who are undergoing prophylactic oophorectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare histologic and molecular alterations in tissue biomarkers of patients at high risk for ovarian cancer treated with celecoxib followed by prophylactic oophorectomy vs prophylactic oophorectomy only.

Secondary

* Compare alterations in gene expression pattern in patients treated with these regimens.

OUTLINE: This is a pilot study. Patients are assigned to 1 of 2 treatment groups.

* Group I: Patients receive oral celecoxib twice daily for 3 months and then undergo prophylactic oophorectomy.
* Group II: Patients undergo immediate prophylactic oophorectomy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk for ovarian cancer and meets criteria for 1 of the following:

  * Family history of at least 2 ovarian** or breast cancers* among the patient and first- or second-degree relatives in the same lineage

    * Multiple primary cancers in the same person may fulfill this requirement
  * Ashkenazi Jewish ethnicity AND 1 first-degree or 2 second-degree relatives with breast* or ovarian** cancer
  * Ashkenazi Jewish ethnicity AND had prior breast cancer*
  * BRCA1/BRCA2 mutation probability > 20% by BRCAPRO
  * Positive for BRCA1 or BRCA2 mutation
  * First- or second-degree relative with a BRCA1/BRCA2 mutation NOTE: *At least 1 breast cancer must be premenopausal (diagnosed at age 50 or under if menopausal status unknown); ductal carcinoma in situ qualifies as breast cancer

NOTE: **In relatives, only ovarian epithelial cancer, fallopian tube cancer, and primary papillary serous cancer qualifies as ovarian cancer

* No prior or concurrent ovarian cancer, including low malignant potential cancers or primary papillary serous carcinoma of the peritoneum

  * No clinical evidence of ovarian cancer by physical examination, CA 125 evaluation, and pelvic ultrasound

PATIENT CHARACTERISTICS:

Age

* 19 and over

Performance status

* GOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,000/mm^3
* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* No hemophilia or other bleeding disorder
* No serious anemia

Hepatic

* Transaminases normal
* Bilirubin normal

Renal

* Creatinine clearance > 80 mL/min OR
* Creatinine < 2.0 mg/dL

Pulmonary

* No emphysema

Other

* Not pregnant or nursing
* No psychiatric or psychological condition that would preclude giving informed consent
* No concurrent untreated malignancy except nonmelanoma skin cancer
* No other medical condition that would preclude blood draws (e.g., chronic infectious disease)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 3 months since prior adjuvant chemotherapy

Endocrine therapy

* Concurrent adjuvant hormonal therapy (e.g., tamoxifen, leuprolide, or goserelin) allowed

Radiotherapy

* More than 3 months since prior adjuvant radiotherapy

Surgery

* More than 3 months since prior intraperitoneal surgery (laparoscopy or laparotomy)
* No prior oophorectomy

Other

* More than 5 years since prior treatment (excluding hormonal therapy) for metastatic malignancy
* No concurrent participation in other ovarian cancer early detection clinical trials

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Alteration in the histologic and molecular alterations in tissue biomarkers between patients at high risk for ovarian cancer treated with Celecoxib and treated without Celecoxib both having prophylactic oophorectomy. | baseline (day of surgery) and 2 years

SECONDARY OUTCOMES:
Alteration in gene expression between group I and group II | from baseline (surgery) to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Partridge, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States